CLINICAL TRIAL: NCT00782587
Title: Phase I Safety and Tolerability Study of Immediate Post-Operative Intravesical Instillation of Chemophase® (Recombinant Human Hyaluronidase in Combination With Mitomycin) in Patients With Non-Muscle-Invasive Bladder Cancer
Brief Title: Study of Immediate Post-Operative Intravesical Instillation of Chemophase® in Patients With Superficial Bladder Cancer
Acronym: IPOP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Jonathan Leff, M.D., Halozyme Therapeutics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZ2-08-01
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Superficial Bladder Cancer
Keywords: Non-Muscle-Invasive Bladder Cancer; Superficial Bladder Cancer; recombinant human hyaluronidase; rHuPH20; Chemophase®; Mitomycin
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Single arm, open label, single dose, intravesical instillation of Chemophase (combination of rHuPH20 and mitomycin) for appropriate superficial bladder cancer patients within 6 hours of TURBT.
  Interventions: Drug: Chemophase

INTERVENTIONS:
Drug: Chemophase — 40 mg mitomycin with 800,000 U rHuPH20 total volume of 40 mL instilled

SUMMARY:
The purpose of this research study is to test the safety and tolerability of an experimental drug, Chemophase, a combination of recombinant human hyaluronidase, (an investigational synthetic enzyme also known as rHuPH20), and mitomycin (MMC) in the treatment of superficial bladder cancer when instilled intravesically immediately after TURBT (transurethral resection of bladder tumor).

DETAILED DESCRIPTION:
Patients will be screened and enrolled prior to undergoing standard of care TURBT for known or suspected Stage Ta, T1 or Tis bladder cancer of any histological grade requiring TURBT and who are believed to be candidates for IPOP intravesical chemotherapy regardless of the need for further intravesical therapy. Within 6 hours after completion of TURBT, patients will be administered a single IPOP intravesical instillation of Chemophase with a one-hour dwell time. At the end of the one-hour dwell time, the patient will be asked to fully void or, if an intravesical catheter has been left in place, the bladder will be fully drained via the catheter. Patients will return at 1 and 2 weeks post instillation for follow up visits for safety and for a cystoscopy at day 85 (per standard of care). Safety and tolerability will be assessed through physical examinations, vital signs, cystoscopy, hematology (CBC), adverse event reporting, and measurements of plasma levels of MMC.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed or suspected (based on cystoscopy) initial presentation or recurrence of Stage Ta, T1, or Tis transitional cell bladder cancer of any histological grade requiring TURBT.
* Patient believed to be a candidate for immediate post-operative chemotherapy regardless of the need for additional intravesical therapy.
* ECOG performance status of Grade 0 or 1.
* Age ≥ 18 years.
* A negative urine or serum pregnancy test (if female of child-bearing potential) within 14 days prior to Day 1/Week 1.
* Acceptable liver function within 14 days prior to Day 1/Week 1 defined as:
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN), and
* AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 2.5 times ULN.
* Acceptable renal function within 14 days prior to Day 1/Week 1 defined as serum creatinine ≤ 1.5 x ULN.
* Acceptable hematologic status within 14 days prior to Day 1/Week 1 defined as:
* Absolute neutrophil count (ANC) ≥ 1,500/dL,
* Platelet count ≥ 100,000/dL, and
* Hemoglobin ≥ 10.0 g/dL.
* Urinalysis showing no clinically significant abnormalities, except those attributable to bladder cancer.
* For men and women of child-producing potential, agreement to use an effective contraceptive method during the study from enrollment until 2 weeks after the administration of study drug.
* Signed, written, IRB-approved informed consent.

Exclusion Criteria:

* Large resected area (estimated total area > 50 cm²) or suspected deep resection, even in the absence of signs of perforation beyond the muscularis propria or ongoing significant bleeding.
* Known or suspected bladder perforation during TURBT.
* Failure to completely resect all cancerous lesions or suspected presence of muscle-invasive cancer (Stage T2 or higher).
* Previous diagnosis or current presence of bladder fibrosis/contracture, or total bladder capacity estimated at cystoscopy or by other means to be < 150 mL.
* Urinary incontinence or severe irritative voiding symptoms such as urgency, frequency, or nocturia of a severity that would compromise the ability of the patient to retain the study drug intravesical instillation for one hour.
* Bladder cancer recurrence less than 3 months after a previous TURBT.
* Major surgery, other than TURBT or diagnostic surgery, within 28 days prior to Day 1/Week 1.
* Known active, uncontrolled bacterial, viral, or fungal infections, including urinary tract infection.
* Any intravesical therapy within 3 months prior to Week 1/Day 1.
* Systemic therapy including radiation therapy, surgery, chemotherapy, or investigational therapy within one month prior to Day 1/Week 1 (two months for nitrosoureas or MMC), unless given as standard treatment for bladder cancer and provided that patient is free of all treatment-related toxicities as of Day 1/Week 1.
* Known infection with HIV.
* Known active infection with hepatitis B or hepatitis C virus.
* Serious disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor (Halozyme).
* History of hypersensitivity or idiosyncratic reaction to, or other contraindication to, MMC.
* Known allergy to bee or vespid venom.
* Known coagulation disorder or bleeding tendency.
* Ongoing treatment with heparin or other anticoagulation therapy, or anticipation of such therapy during the treatment period in this study.
* Unwillingness or inability to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of immediate post-operative instillation of Chemophase. | Day 1 instillation, and weeks 1, 2, and 12

SECONDARY OUTCOMES:
Assess plasma levels of mitomycin (MMC) after IPOP intravesical instillation. | Hours 1, 2 and 3 post-instillation

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lamm, M.D., Principal Investigator — BCG Oncology, PC
Locations (5):
- United States (5):
  - BCG Oncology, PC, Phoenix, Arizona
  - Advanced Urology Medical Center, Anaheim, California
  - Medresearch, La Mesa, California
  - Malcolm Randall Veterans Administration, Gainesville, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida